CLINICAL TRIAL: NCT05119439
Title: An Outpatient Medical Abortion Regimen With Mifepristone and Two Doses of Misoprostol at 71-77 and 78-84 Days of Pregnancy
Brief Title: Mifepristone and Two Doses of Misoprostol for Abortion at 11&12 Weeks
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment
Sponsor: Gynuity Health Projects (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1050
Record Dates: First submitted 2021-11-05; First posted 2021-11-15 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Medical Abortion
Keywords: mifepristone; misoprostol; first trimester; abortion
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 71-77 days of gestational age (No Intervention): Pregnant people whose pregnancies are estimated to have a gestational age of 71-77 days. (Participants in this arm receive the standard of care for medical termination of pregnancy in the stated gestational age range).
- 78-84 days of gestational age (Experimental): Pregnant people whose pregnancies are estimated to have a gestational age of 78-84 days.
  Interventions: Drug: Mifepristone + 2 doses of misoprostol 800 mcg

INTERVENTIONS:
Drug: Mifepristone + 2 doses of misoprostol 800 mcg — Will use a mifepristone-misoprostol regimen of: 200 mg mifepristone followed in 24-48 hours by a first dose of 800 µg misoprostol buccally and then in another 4 hours by a second dose of 800 µg misoprostol buccally. For buccal administration of misoprostol, participants will place 2 misoprostol tablets in each cheek and hold them for 20-30 minutes, after which they will swallow any remnants.
  Arms: 78-84 days of gestational age

SUMMARY:
This study seeks to evaluate the efficacy, side effect profile and acceptability of a medical abortion regimen with mifepristone and two doses of 800 mcg misoprostol buccally at 71-77 and 78-84 days of gestation to further expand the evidence base for the most effective regimens in the late first trimester of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Seeking medical abortion services at one of the enrolling clinics
* Have an intrauterine pregnancy 71-77 days of gestation or 78-84 days
* Meet standard eligibility criteria for medical abortion
* Be able to return to clinic for in-person follow up
* Speak/read/write English or Spanish
* Have access to a mobile phone with texting capability
* Be in general good health
* Be willing and able to sign consent forms
* Agree to comply with the study procedures and follow up.

Exclusion Criteria:

* Not eligible to consent on their own to being in a study (Age criteria may vary by site according to state law.)
* With known allergies or other contraindications to mifepristone or misoprostol
* Desiring to start depot medroxyprogesterone acetate (DMPA) as contraception method immediately because of potential interaction with mifepristone. Those who wish to wait until abortion completion to start DMPA will be eligible for enrollment.

Ages: 11 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Efficacy as determined by the proportion of successful abortions without aspiration or D&E for any reason | 7-36 days after initial visit
  Proportion of women who achieve complete abortion with medication only and without aspiration or D&E

SECONDARY OUTCOMES:
Proportion of participants who report each individual side effect | 7-14 days after initial visit
  Side effects include diarrhea, nausea, vomiting, fever, chills
Proportion of complications experienced by participants that warrant visits to emergency room and/or hospitalization | 7-14 days after initial visit
  Complications could include abnormal bleeding, severe pain, retained tissue
Proportion of participants who determine method acceptable | 7-36 days after initial visit
  Overall acceptability, time to complete abortion, bleeding, side effects, pain

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (6):
- United States (6):
  - University of Hawaii, Hilo, Hawaii
  - University of Hawaii, Honolulu, Hawaii
  - Planned Parenthood North Central States, Saint Paul, Minnesota
  - Philadelphia Women's Center, Philadelphia, Pennsylvania
  - Planned Parenthood Great Northwest, Hawai'i, Alaska, Indiana, Kentucky, Federal Way, Washington
  - Planned Parenthood Great Northwest, Hawai'i, Alaska, Indiana, Kentucky, Tacoma, Washington